CLINICAL TRIAL: NCT04327479
Title: Characterization of Cardiovascular Diseases and Risk Factors in Patients With Suspected SARS-CoV2/Covid-19 Infection
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: 20-9213-BO
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; SARS
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessment of cardiovascular diseases and cardiovascular risk factors — At inclusion, patients will be screened for pre-existing cardiovascular diseases and cardiovascular risk factors, as well as medication.

SUMMARY:
The Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infects host-cells via ACE2-receptors, which leads to pneumonia (COVID-19) but also can lead to myocarditis (acute myocardial injury) and chronic damage to the cardiovascular system. Therefore, cardiovascular protection may be necessary when treating patients with COVID-19 infection. This may especially be necessary in patients with cardiovascular diseases, risk factors, and co-medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected SARS-CoV2/Covid-19 infection

Exclusion Criteria:

* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will include consecutive patients, tested for suspected SARS-CoV2/Covid-19 infection at the University Hospital Essen
Sampling Method: Probability Sample
Enrollment: 728 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | During 1 year follow-up
  mortality of any cause

SECONDARY OUTCOMES:
30-day mortality | Within 30 days after inclusion
  mortality of any cause
Major adverse cardiovascular events | During 1 year follow-up
  Myocardial infarction, stroke, or CV death

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, MD, Principal Investigator — University Hospital Essen, Deparment of Cardiology and Vascular Medicine
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Will be made available upon request

REFERENCES:
- [Derived] Mahabadi AA, Mincu R, Dykun I, Michel L, Kung A, Witzke O, Kill C, Buer J, Rassaf T, Totzeck M. Frequency and prognosis of CVD and myocardial injury in patients presenting with suspected COVID-19 - The CoV-COR registry. Int J Cardiol Heart Vasc. 2023 Apr;45:101184. doi: 10.1016/j.ijcha.2023.101184. Epub 2023 Feb 6. PMID 36776683